CLINICAL TRIAL: NCT07328529
Title: Safety, Tolerability, and Efficacy of SRX246, a Vasopressin 1a Receptor Antagonist, in Aggressive Participants With Fragile X Syndrome
Brief Title: Inhibition of Aggressive Behavior in Participants With Fragile X Syndrome
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Azevan Pharmaceuticals (Industry)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AVN014; CDMRP-PR240390 (Other Grant/Funding Number: Congressionally Directed Medical Research Programs (CDMRP))
Record Dates: First submitted 2026-01-07; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Aggressive Behavior in Fragile X Syndome
Keywords: Fragile X Syndrome; SRX246; vasopressin 1a; irritability; agitation; aggression; self-injury
MeSH Terms: conditions — Fragile X Syndrome; Psychomotor Agitation; Aggression; Self-Injurious Behavior | interventions — SRX246

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SRX246 (Experimental): SRX246 will be provided as 120mg capsule to be taken orally, twice per day, once in the morning and once in the evening.
  Interventions: Drug: SRX246
- Placebo (Placebo Comparator): Placebo will be provided as a matching capsule to be taken orally, twice per day, once in the morning and once in the evening.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SRX246 — SRX246 120mg capsules for oral administration
  Arms: SRX246
Drug: Placebo — Placebo capsules for oral administration
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if drug SRX246 works to treat irritability, agitation, aggression and self-injury (IAAS) behaviors in adult males with Fragile X Syndrome (FXS). It will also learn about the safety of drug SRX246. The main questions it aims to answer are:

* Does drug SRX246 lower the number of times participants experience IAAS behaviors?
* What medical problems do participants have when taking drug SRX246? Researchers will compare drug SRX246 to a placebo (a look-alike substance that contains no drug) to see if drug SRX246 works to treat IAAS behaviors.

Participants will:

* Take drug SRX246 or a placebo every day for up to 8 months
* Have weekly checkups by phone or video to answer study questions
* Have periodically scheduled home visits by nurses to conduct medical check-ups and tests
* Keep a diary of their symptoms

ELIGIBILITY:
Inclusion Criteria:

* Biological male, age 18 to 45 years inclusive
* Molecular genetic confirmation of the full Fragile X messenger ribonucleoprotein mutation (≥200 CGG repetitions)
* IAAS symptoms leading to a CGI-S score for Disruptive Behavior of 5 or more
* Reported history of aggression based on the CMAI-Agg subscale (average score >22) and an average associated disruptiveness scale of at least 3.
* IQ < 70
* Stable medication doses for the last month
* Has a caregiver who lives with or spends extensive time with the participant most days and can report behavioral symptoms
* Must be able to swallow study drug capsules whole

Exclusion Criteria:

* Medical condition contraindicating study participation
* SGPT and SGOT values 2 or more times the upper limit of normal
* History of psychosis
* Suicidal behavior

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Aberrant Behavior Checklist | Over an 8 month period
  The Aberrant Behavior Checklist-Community Edition (ABC-C) Irritability subscale - Caregiver rated and then scored using the using the FXS-specific factoring system (ABCFX). Responses will be rated using a scale ranging from 0=not a problem to 3=severe problem.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of California, Davis, MIND Institute, Sacramento, California
  - Rush University Medical Center, Chicago, Illinois
  - Cincinnati Children's Hospital, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Yes